CLINICAL TRIAL: NCT00590798
Title: Star-Close Early Ambulation Trial
Acronym: STRUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ernest Mazzaferri (Other)
Responsible Party: Sponsor-Investigator, Ernest Mazzaferri, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STRUT
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Cardiovascular Disease
Keywords: Cardiac Catheterization; Walk; Heart Catheterization; Coronary Disease; Heart Disease; Coronary Artery Disease
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Coronary Artery Disease | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients are asked to walk within 30 minutes after implantation of the Star- Close vascular closure system.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Walking — Patient will walk within 30 minutes of vascular closure system procedure

SUMMARY:
To confirm that patients who receive the Star-Close vascular closure system (VCS) can safely ambulate within 30 minutes of catheterization.

DETAILED DESCRIPTION:
To confirm that patients who receive the Star-Close vascular closure system (VCS) after diagnostic cardiac catheterization can safely ambulate within 30 minutes of catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to for an outpatient left heart catheterization
* Catheterization through the femoral artery
* Able to ambulate at least 20 feet
* Able to receive the Star-Close Vascular Closure System
* Be a candidate for hospital discharge following catheterization

Exclusion Criteria:

* Known peripheral arterial disease
* Blood pressure greater than 180/110
* Pregnant or lactating
* Anemic or low blood count
* Blood thinning medication within 5 days before catheterization
* Unable to walk 20 feet with out rest
* Complications during catheterization procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Occurrence or absence of adverse outcomes after ambulation within 30 minutes of cardiac catheterization | 7 days post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Earnest L Mazzaferri Jr, MD, Principal Investigator — The Ohio State University Medical Center, Division of Cardiovascular Medicine
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States